CLINICAL TRIAL: NCT06497777
Title: The Application of DNA Nanomachines for Detecting microRNA in Blood for the Diagnosis of Pancreatic Cancer.
Brief Title: The Application of DNA Nanomachines for Detecting microRNA in Blood for the Diagnosis of Pancreatic Cancer. Diagnosis of Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202405082RINB
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Adenocarcinoma; MicroRNA
Keywords: MicroRNA; Pancreas Adenocarcinoma
MeSH Terms: interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic adenocarcinoma: Pancreatic adenocarcinoma which are proven by pathology, before initiation of anti-cancer treatment.
  Interventions: Genetic: MicroRNA (mir-642b-3p)
- Healthy control: People who do not have pancreatic disease.

INTERVENTIONS:
Genetic: MicroRNA (mir-642b-3p) — A circulating microRNA in the blood of pancreatic cancer patients.
  Groups: Pancreatic adenocarcinoma

SUMMARY:
Previous research has shown that microRNAs in the blood can serve as biomarkers for early pancreatic cancer, with potential applications including detection, differential diagnosis, and prognosis prediction of pancreatic cancer. The current primary method for detecting microRNAs is RT-qPCR, but this process requires repeated temperature cycling, which demands high precision from the equipment. As an alternative, isothermal nucleic acid amplification technology does not require expensive temperature control instruments. Our research team has developed various isothermal nucleic acid amplification strategies for microRNA sensing platforms, applied to biological sample detection. This study combines the circular strand displacement amplification strategy with DNA nanomachines to develop a fluorescence sensing platform that performs dual signal amplification at a constant temperature. It is designed to detect pancreatic cancer-related microRNAs, exploring its role and potential applications in the diagnosis of pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic ductal adenocarcinoma
* Proven by pathology
* Patients who have not received anti-cancer therapies

Exclusion Criteria:

* Less than 20 years old
* Unable to provide inform and consent
* Patients who have active malignancy other than pancreatic adenocarcinoma
* Patients who have had pancreatic cancer whose anti-cancer therapies are completed or undergoing
* Life expectancy less than 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic ductal adenocarcinoma which are proven by pathology.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-06 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Ratio of the target microRNA in patients with and without pancreatic adenocarcinoma. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan